CLINICAL TRIAL: NCT03411109
Title: Efficacy and Outcomes of Intrathecal Analgesia As Part of an Enhanced Recovery Pathway in Colon and Rectal Surgical Patients
Brief Title: Outcomes of Intrathecal Analgesia in Colorectal Surgery
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Adam K. Jacob, Principal Investigator, Mayo Clinic
Other Study IDs: 13-007936
Record Dates: First submitted 2018-01-19; First posted 2018-01-25 (Actual); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Surgery
Keywords: intrathecal analgesia; colorectal; enhanced recovery
MeSH Terms: interventions — Hydromorphone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Opioid Only Intrathecal
  Interventions: Drug: Hydromorphone Hydrochloride
- Opioid + Local Anesthetic Intrathecal
  Interventions: Drug: Hydromorphone Hydrochloride

INTERVENTIONS:
Drug: Hydromorphone Hydrochloride — All intrathecal injections were performed preoperatively using a 22g or 25 g Whitacre or 24g Sprotte spinal needle. The IA regimen, medication(s) and dose(s), was at the discretion of the attending anesthesiologist, and consisted of one of the following regimens: (1) hydromorphone + local anesthetic (IA-L), or (2) hydromorphone only (IA-O). In patients receiving IA, no other interventional locoregional analgesic techniques (such as rectus sheath blocks or transversus abdominis plane blocks) were utilized.

SUMMARY:
Multimodal analgesia, sometimes including intrathecal analgesia (IA), is essential in any enhanced recovery pathway (ERP). This study aimed to evaluate the safety, feasibility, and optimal IA regimen in colorectal surgical patients.

ELIGIBILITY:
Inclusion Criteria:

* All adult colorectal patients from October 2012 through December 2013 in which patients received single-injection IA as part of a multimodal analgesic strategy for ERP.
* Undergoing an elective colorectal operation (minimally invasive or open)

Exclusion Criteria:

* Patients aged < 18 years
* American Society of Anesthesiologists (ASA) 5 and 6 classification
* pregnancy
* failure to provide research authorization.
* emergent operations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients receiving colorectal surgical care at a tertiary care, academic institution.
Sampling Method: Non-Probability Sample
Enrollment: 601 (Actual)
Dates: Start 2012-10-01 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2013-12-31 (Actual)

PRIMARY OUTCOMES:
Time to return of bowel function | post resection, approximately up to 48 hours
  Time to return of bowel function is defined by the presence of flatus and a bowel movement

CONTACTS AND LOCATIONS:
Overall Officials: Adam Jacob, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Merchea A, Lovely JK, Jacob AK, Colibaseanu DT, Kelley SR, Mathis KL, Spears GM, Huebner M, Larson DW. Efficacy and Outcomes of Intrathecal Analgesia as Part of an Enhanced Recovery Pathway in Colon and Rectal Surgical Patients. Surg Res Pract. 2018 Mar 1;2018:8174579. doi: 10.1155/2018/8174579. eCollection 2018. PMID 29687077